CLINICAL TRIAL: NCT01971463
Title: Optical Measurement of Cerebral Blood Flow Response After Ischemic Stroke
Brief Title: Bolus of Saline in Stroke
Acronym: BOSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 818577
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal Saline (Experimental): intravenous administration of 500cc of 0.9% NaCl over 30 minutes
  Interventions: Other: Normal saline

INTERVENTIONS:
Other: Normal saline — intravenous administration of 500cc of 0.9% NaCl over 30 minutes

SUMMARY:
This study is a non-randomized, Phase 2 clinical trial designed to assess optical cerebral blood flow (CBF) response to bolus normal saline. Subjects will have had an ischemic stroke within 96 hours of enrollment. The study intervention will be a one hour monitoring session. There will be a 15 minute baseline measurement period, followed by intravenous administration of 500cc of 0.9% NaCl over 30 minutes, and finally 15 minutes of monitoring post-bolus. All study measurements will cease after 1 hour. Subjects will be followed during their hospitalization for 7 days or until discharge, whichever is sooner, to monitor for adverse events and to collect clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute ischemic stroke in the territory of the anterior, middle, or posterior cerebral artery territory on either side of the brain
* Study intervention can be initiated within 96 hours of symptom onset
* Willingness and ability to sign informed consent by patient or legally acceptable surrogate decision-maker

Exclusion Criteria:

* Infarct limited to the brainstem and/or cerebellum with no involvement of the cerebral hemispheres
* Bi-hemispheric infarction or acute infarct in the contra-lateral hemisphere within the past 30 days
* Symptoms of active congestive heart failure (dyspnea, orthopnea, increased oxygen requirement)
* Exacerbation of congestive heart failure, requiring hospitalization, within the past 30 days or severe systolic dysfunction with a known ejection fraction <20%
* End stage renal disease requiring hemodialysis or a creatinine clearance <20 ml/min/1.73 m2
* Hemicraniectomy or other skull defect that would interfere with monitoring
* Pregnant women are excluded. Women of child-bearing age must have a negative pregnancy test prior to enrollment
* Participation in another clinical trial
* Any other illness or condition that the investigator feels would pose a hazard to the subject from participation in the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline
Started | 81
Completed | 81
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 81 subjects enrolled. A technical advancement in DCS fiber optic probe design increased signal-to-noise ratio occurred after the first 8 subjects; these subjects were excluded because their data was not comparable to later subjects. 5 subjects who failed to complete the monitoring session and 11 subjects were excluded due to poor data quality.
Arm/Group | Normal Saline
Number analyzed (Participants) | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [53 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Time from symptom onset [Median (Inter-Quartile Range); unit: hours] | 66 [49 to 83]
NIH Stroke Scale [Median (Inter-Quartile Range); unit: units on a scale] — The National Institutes of Health Stroke Scale (NIHSS) is a measure of stroke severity, ranging from 0-42, with 0 representing no neurologic deficit and 42 representing severe neurologic impairment.
  units on a scale | 2 [1 to 7]

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Change in Optical Cerebral Blood Flow (oCBF) During Bolus Normal Saline Compared to Baseline, as Measured by Diffuse Correlation Spectroscopy (DCS).
Description: Ipsilesional hemisphere
Time Frame: 30 minutes after completion of saline bolus
Measure: Median (Inter-Quartile Range); unit: percent change from baseline flow
Arm/Group | Normal Saline
Number analyzed (Participants) | 57
percent change from baseline flow | 17 [-2.0 to 43.1]

2. Primary Outcome: The Percentage of Change in Optical Cerebral Blood Flow (oCBF) During Bolus Normal Saline Compared to Baseline, as Measured by Diffuse Correlation Spectroscopy (DCS).
Description: contralesional hemisphere
Time Frame: 30 minutes after completion of saline bolus
Measure: Median (Inter-Quartile Range); unit: percent change from baseline flow
Arm/Group | Normal Saline
Number analyzed (Participants) | 57
percent change from baseline flow | 13.3 [-4.3 to 36.0]
Statistical Analysis 1: Comparison: Normal Saline; Change in oCBF from baseline to post-bolus, ipsilesional hemisphere; Test type: Superiority; p < 0.05, Wilcoxon signed rank
Statistical Analysis 2: Comparison: Normal Saline; Test type: Superiority — Mixed effects regression, modeling the interaction term for time x normal saline bolus in the ipsilesional hemisphere; p < 0.001, Mixed Models Analysis; Slope = 0.05, 95% CI 2-sided [0.03 to 0.07]

ADVERSE EVENTS:
Arm/Group | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 3/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=81)
IV infiltration (Vascular disorders) | 1 (1)
Elevated systolic blood pressure (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) — Subject was in atrial fibrillation at start of monitoring session, developed tachycardia during monitoring due to rapid ventricular response

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No